CLINICAL TRIAL: NCT07314593
Title: Effectiveness of Cod-Derived Omega Oil Enriched With Free Fatty Acids Against the Common Cold and Other Respiratory Infections in Healthy Icelandic Adults During the Influenza Season
Brief Title: Omega-Cold Supplementation With Free Fatty Acids for the Prevention of Respiratory Infections in Adults.
Acronym: OmegaCold FFA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Landspitali University Hospital (Other)
Collaborators: Matis ohf. (Unknown); Lipid Pharmaceuticals ehf. (Unknown)
Responsible Party: Principal Investigator, Magnus Gottfredsson, Principal Investigator, Landspitali University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 62870 - Omega Cold FFA
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Infections
Keywords: Free Fatty Acids; Common Cold; respiratory infections; Omega-3; Influenza; COVID-19
MeSH Terms: conditions — Respiratory Tract Infections; Common Cold; Influenza, Human; COVID-19 | interventions — Docosahexaenoic Acids; Fatty Acids, Nonesterified

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 oil with Free Fatty Acids (Experimental): Omega-3 oil enriched with Free Fatty Acids (2%)
  Interventions: Dietary Supplement: Omega-3 oil with 2% Free Fatty Acids
- Placebo (Placebo Comparator): Vegetable oil as a placebo
  Interventions: Dietary Supplement: Vegatable oil

INTERVENTIONS:
Dietary Supplement: Omega-3 oil with 2% Free Fatty Acids — Omega-3 oil enriched with Free Fatty Acids (2%) for oral intake
  Arms: Omega-3 oil with Free Fatty Acids
Dietary Supplement: Vegatable oil — Vegetable oil as placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate whether fish oil containing free fatty acids affects people's susceptibility to viral infections such as colds, influenza, and COVID-19, as well as the course of these illnesses. Omega Cold is purified fish oil with 2% added free fatty acids, making it similar in that respect to less-purified fish oils. Participants aged 18-80 in generally good health will be recruited through Matís' consumer mailing list and social media advertisements. A total of 400 participants are planned: 100 in the winter of 2025-2026 and 300 in the winter of 2026-2027. Participants will be randomly assigned to two equal groups. One group will take Omega Cold orally twice a day for four months, while the other receives a placebo (vegetable oil) taken in the same way. They will not be asked to change any other habits. All participants will report weekly on their health and any cold or flu symptoms during the time they take the oil, using short questionnaires. The study is scheduled to begin in December 2025, when the oil will be sent to participants.

DETAILED DESCRIPTION:
The purpose of the Omega Cold fish oil study is to determine whether fish oil enriched with free fatty acids affects people's susceptibility to viral infections, such as colds, flu or COVID, and the illnesses caused by such infections.

Free fatty acids are present in untreated fish oil. However, the fish oil most commonly on the market today has been purified of free fatty acids. Omega Cold fish oil is purified fish oil with added free fatty acids in 2% concentration. This study is the first step in investigating whether fish oil with free fatty acids affects how often people get sick from viral infections, and whether consuming the fish oil affects the progression of the illness.

Participants in the study are recruited by sending an email to Matís' consumer list and through advertisements on social media. The conditions for participation are to be between the ages of 18-80 and in generally good health. The aim is for 400 people to participate in the study - 100 in the winter of 2025 - 2026 and 300 in the winter of 2026 - 2027.

The participants will be divided into two equal groups. One group will receive Omega Cold fish oil to take twice a day for four months. The other group is a placebo group and will receive vegetable oil to take in the same way. Participants will not be asked to change anything else in their consumption or behavior. All participants will be asked to record information about their health with regard to cold and flu symptoms weekly during the time they take the oil using short questionnaires.

ELIGIBILITY:
Inclusion Criteria: To be in general good health, be between 18 to 80 years of age and be willing and able to take fish oil orally.

-

Exclusion Criteria: Younger than 18 years and older than 80 years.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Frequency, duration and severity of respiratory infections | Four months
  Participants will complete a short weekly questionnaire reporting any respiratory infection symptoms they experienced in the past seven days. If symptoms are present, they will be asked to provide additional details, including the type of symptoms, their duration, and their severity rated on numerical scales.

CONTACTS AND LOCATIONS:
Overall Officials: Magnús Gottfreðsson, MD, PhD, Principal Investigator — Landspitali, University of Iceland

IPD SHARING:
Plan to Share IPD: No